CLINICAL TRIAL: NCT01162941
Title: Efficacy of Helicobacter Pylori Eradication, Anti-D and Danazol Combination in Steroid Dependant or Refractory Immune Thrombocytopenia (ITP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-019
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Thrombocytopenia | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Steroid dependant ITP (Experimental): more than 10 mg of prednisolone per day is required to maintain a platelet count above 20X109/L (minimum follow up duration: 3 months after diagnosis)
  Interventions: Other: Steroid refractory ITP

INTERVENTIONS:
Other: Steroid refractory ITP — a platelet count less than 20X109/L despite of treatment with full dose of steroid (prednisolone 1mg/kg for at least 4 weeks)
  Other Names: prednisolone 1mg/kg

SUMMARY:
Proportion who would avoid splenectomy at 6 months of follow up

DETAILED DESCRIPTION:
1. If urea breath test (+); omeprazole 20mg bid, amoxicillin 1000mg bid and clarithromycin 500mg bid for 1 week.

   Second line Helicobacter pylori eradication will be permitted after failure of first line treatment.
2. Anti-D Anti-Ro 50 μg/kg IV for 2 days (D1, 2)
3. Danazol maintenance (from D1): Danazol will be continued at least 3 months. The dose of danazol can be reduced according to the adverse effects, especially in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* 1.ITP is defined by

  * (a) a true thrombocytopenia on blood smear, (b) adequate megakaryopoiesis on bone marrow examination, (c) the absence of clinically apparent associated conditions or cause of thrombocytopenia
* 2.Steroid dependant ITP: more than 10 mg of prednisolone per day is required to maintain a platelet count above 20X109/L (minimum follow up duration: 3 months after diagnosis)
* 3.Steroid refractory ITP: a platelet count less than 20X109/L despite of treatment with full dose of steroid (prednisolone 1mg/kg for at least 4 weeks)
* 4.18 years old or more

Exclusion Criteria:

* 1.Patients who have a cause of thrombocytopenia such as HIV infection, lymphoproliferative disease, liver disease, definite SLE or drug
* 2.Pregnancy
* 3.Splectomized patients
* 4.Rh- blood type
* 5.Hemoglobin < 10g/dL
* 6.Known hypersensitivity to immunoglobulins
* 7.A positive direct antiglobulin test
* 8.Clinically relevant hepatic or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-07 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Proportion who would avoid splenectomy at 6 months of follow up | 2years
  Proportion who would avoid splenectomy at 6 months of follow up

SECONDARY OUTCOMES:
SR,IR | 2years
  Sustained response (platelet count that remained above 30X109/L or 2 folds of initial platelet count at 6 months of follow up) Initial response (an increase in the platelet count of at least 10X109/L or a platelet count of more than 30X109/L by day 7 after the initiation of treatment) Changes of platelet counts Safety of treatment Response rate of HP infected patients Decrement of steroid dose Predictors of response

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hee Lee, professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Asanbyeongwon-gil, Songpa-gu, South Korea

REFERENCES:
- See also: Efficacy of Helicobacter pylori eradication, anti-D and danazol combination in steroid dependant or refractory immune thrombocytopenia (ITP) — http://www.google.co.kr